CLINICAL TRIAL: NCT05569148
Title: A Phase IIIb, Open-Label, Single-Arm Study in Patients With Neovascular Age-Related Macular Degeneration or Diabetic Macular Edema to Evaluate the Safety of the 6-mg Faricimab Prefilled Syringe
Brief Title: A Study in Patients With Neovascular Age-Related Macular Degeneration or Diabetic Macular Edema to Evaluate the Safety of the Faricimab Prefilled Syringe
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GR43742
Record Dates: First submitted 2022-10-04; First posted 2022-10-06 (Actual); Results first posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-09

CONDITIONS: Neovascular Age-related Macular Degeneration; Diabetic Macular Edema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Faricimab PFS Configuration (Experimental)
  Interventions: Combination Product: Faricimab PFS Configuration

INTERVENTIONS:
Combination Product: Faricimab PFS Configuration — Participants will receive a single intravitreal (IVT) injection of the 6-milligram (mg) faricimab dose formulation delivered via prefilled syringe (PFS) with a co-packaged injection filter needle.
  Other Names: VABYSMO™; RO6867461; RG7716

SUMMARY:
This Phase IIIb, single-arm, open-label multicenter clinical in-use study in patients with neovascular age-related macular degeneration (nAMD) or diabetic macular edema (DME) is designed to assess the ability of the intended users, healthcare providers (HCPs), to follow the Instructions for Use to perform an intravitreal (IVT) injection using the 6-milligram (mg) faricimab prefilled syringe (PFS) configuration per the intended use. Any adverse events occurring during the 7-day study reporting period will be summarized.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to comply with clinic visits and study-related procedures
* For female patients of childbearing potential: agree to remain abstinent (refrain from heterosexual intercourse) or use contraception, and agree to refrain from donating eggs, as defined in the protocol
* Confirmed diagnosis of neovascular age-related macular degeneration (nAMD; any subtype) or diabetic macular edema (DME) in one or both eyes by the study site investigator (only one eye will be selected as the study eye, as determined by the retina specialist) with onset at any time prior to study start
* Study eye is deemed to be indicated for faricimab intravitreal (IVT) treatment at the discretion of the retina specialist
* Hstorical optical coherence tomography (OCT) data available for the study eye within 30 days prior to Day 1

Exclusion Criteria:

* Pregnancy or breastfeeding, or intention to become pregnant during the study or within 3 months after the final dose of faricimab
* Requirement on Day 1 for continuous use of any medications and treatments considered prohibited therapy per the protocol
* Participation in an investigational trial that involves treatment with any drug or device (with the exception of vitamins and minerals) within 3 months prior to Day 1
* Stroke (cerebral vascular accident) or myocardial infarction within 6 months prior to Day 1
* History of a severe allergic reaction or anaphylactic reaction to a biologic agent or known hypersensitivity to any component of the faricimab prefilled syringe injection, study-related procedure preparations, or any of the anesthetic and antimicrobial preparations used by a participant during the study
* History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a condition that contraindicates the use of faricimab or renders the patient at high risk for treatment complications in the opinion of the investigator
* Uncontrolled hypertension (systolic blood pressure >180 mmHg and/or diastolic blood pressure >100 mmHg while a patient is at rest)
* Systemic treatment for suspected or active systemic infection on Day 1
* Legally blind in the study eye on Day 1 (legal blindness: Best-corrected visual acuity [BCVA] of 20/200 or less)
* History of or any current clinically relevant intraocular inflammation or ocular inflammatory reaction (any grading from trace and greater is excluded), including non-infectious uveitis or infectious uveitis, or sterile inflammatory reaction after previous IVT injections with any agent in either eye
* Suspected or active ocular or periocular infection in either eye on Day 1
* History of or any current indication of excessive bleeding and recurrent hemorrhages, including any prior excessive intraocular or subconjunctival bleeding or hemorrhages after IVT injection or intraocular procedures in either eye
* Uncontrolled glaucoma in the study eye
* Treatment with any IVT injection in the study eye within the 27 days prior to Day 1
* Any invasive intraocular surgery, prior long-acting therapeutic agent, or ocular drug release device implantation (approved or investigational) in the study eye at any time during the 3 months prior to Day 1
* Treatment with panretinal photocoagulation, laser retinopexy or macular (focal, grid, or micropulse) laser in the study eye within one month prior to Day 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2022-10-17 (Actual); Primary Completion 2022-11-10 (Actual); Study Completion 2022-11-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (3):
- United States (3):
  - Barnet Dulaney Perkins Eye Center, Mesa, Arizona
  - Associated Retina Consultants, Phoenix, Arizona
  - Retinal Consultants of Arizona, Phoenix, Arizona

IPD SHARING:
Plan to Share IPD: No
Qualified researchers may request access to individual patient level data through the request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/).
  For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

REFERENCES:
- [Derived] Barakat MR, Kwong HM Jr, Marcon G, O'Leary OE, Paris LP, Schneider P, Tang Y, Graff JM. Human Factors Studies to Assess the Usability of the Faricimab Prefilled Syringe. Clin Ophthalmol. 2025 Feb 6;19:395-406. doi: 10.2147/OPTH.S503060. eCollection 2025. PMID 39931677

RESULTS

PARTICIPANT FLOW:
Groups:
- Faricimab PFS Configuration: Healthcare providers (HCP) prepared and administered a single intravitreal (IVT) injection of the 6-milligram (mg) faricimab dose formulation to each patient via prefilled syringe (PFS) with a co-packaged injection filter needle on Day 1.
Period: Overall Study
Arm/Group | Faricimab PFS Configuration
Started | 35
Completed | 35
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All enrolled patients
Arm/Group | Faricimab PFS Configuration
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: Years] | 74.7 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 32
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 33
  More than one race | 0
  Unknown or Not Reported | 1
Underlying Condition in Study Eye [Count of Participants; unit: Participants] — DME = diabetic macular edema; nAMD = neovascular age-related macular degeneration (nAMD)
  Participants
    DME Only | 12
    nAMD Only | 22
    Both DME and nAMD | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Injection Procedures With Successful Completions on Critical Tasks Performed by Healthcare Providers in the Use of the Faricimab Prefilled Syringe Configuration
Description: Thirteen healthcare providers (HCP; seven retina specialists and six assistants) across three sites participated in the study, and they worked mostly in pairs to administer a single intravitreal (IVT) injection of 6-mg faricimab to each of the 35 patients using the prefilled syringe (PFS). For each IVT injection, two Human Factors (HF) observers were positioned such that they could clearly observe the entire preparation and administration process. Each HCP team (i.e., retina specialist alone or retina specialist with assistant, as per local procedure) were asked to perform all preparation and administration steps in view of the HF observers. Critical tasks were observed by the HF observers who documented HCP performance using an assessment checklist. A successful task completion for each critical task was defined as normal use without use error, and the percentages of successful completions are calculated out of the total 35 PFS IVT injections administered.
Time Frame: Day 1
Population: The target population included all 35 enrolled patients. Thirteen HCPs (7 retina specialists and 6 assistants) performed tasks to prepare and administer a single faricimab PFS IVT injection to each of the 35 patients. Certain critical tasks could only be performed by the retina specialists.
Measure: Number; unit: Percentage of injection procedures
Units Other Than Participants: Injection Procedures
Arm/Group | Faricimab PFS Configuration
Number analyzed (Participants) | 35
Number analyzed (Injection Procedures) | 35
Percentage of injection procedures
  Open Folding Box | 100
  Remove Leaflet and Tray with Syringe from Folding Box | 100
  Remove Supplied Injection Filter Needle from Folding Box | 100
  Peel Lid off the Tray | 100
  Aseptically Remove Syringe from Tray | 100
  Split Open Pouch | 100
  Aseptically Remove Injection Filter Needle | 100
  Remove Syringe Tip Cap | 100
  Aseptically Attach Supplied Injection Filter Needle Onto Syringe Luer Connector | 100
  Remove Injection Filter Needle Cap | 100
  Hold Syringe Upright | 100
  If Air Bubbles are Present, Tap to Force Air Bubbles to the Top of the Syringe | 100
  Slowly Push the Plunger to Align the Stopper to the Syringe 0.05 mL Dose Mark | 100
  Insert Injection Filter Needle at the Injection Site | 100
  Inject Slowly Until Stopper Reaches the End of the Syringe Barrel to Deliver the Volume of 0.05 mL | 100
  Remove Injection Filter Needle from the Injection Site | 100
  Dispose of Used Syringe with Uncapped Needle in a Sharps Disposal Container | 100

2. Primary Outcome: Percentage of Injection Procedures With Use Errors on Critical Tasks Performed by Healthcare Providers in the Use of the Faricimab Prefilled Syringe Configuration
Description: Thirteen healthcare providers (HCP) across 3 sites participated in the study, and they worked mostly in pairs to administer a single intravitreal (IVT) injection of 6-mg faricimab to each of the 35 patients using the prefilled syringe (PFS). For each IVT injection, two Human Factors (HF) observers were positioned such that they could clearly observe the entire preparation and administration process. Each HCP team (i.e., retina specialist alone or retina specialist with assistant, as per local procedure) were asked to perform all preparation and administration steps in view of the HF observers. Critical tasks were observed by the HF observers who documented HCP performance using an assessment checklist. A use error was defined as user action or lack of user action while using the medical device that leads to a different result than that intended by the manufacturer or expected by the user. The percentages of use errors are calculated out of the total 35 PFS IVT injections administered.
Time Frame: Day 1
Population: as for outcome 1
Measure: Number; unit: Percentage of injection procedures
Units Other Than Participants: Injection Procedures
Arm/Group | Faricimab PFS Configuration
Number analyzed (Participants) | 35
Number analyzed (Injection Procedures) | 35
Percentage of injection procedures | 0

ADVERSE EVENTS:
Time Frame: From Day 1 to Day 7
Arm/Group | Faricimab PFS Configuration
All-Cause Mortality (participants affected / at risk) | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35
Other Adverse Events (participants affected / at risk) | 1/35
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Faricimab PFS Configuration (N=35)
Eye irritation (Eye disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study being conducted under this agreement is part of the overall study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the study, but only after the first publication or presentation that involves the overall study. The Sponsor may request that confidential information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol (2022-06-29): https://cdn.clinicaltrials.gov/large-docs/48/NCT05569148/Prot_001.pdf